CLINICAL TRIAL: NCT04106674
Title: Conservative Versus Operative Treatment of Two - Part Proximal Humerus Fractures
Brief Title: Two- Part Proximal Humerus - Conservative vs Operative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Hendrik Frolich Fuglesang, Consultant, Head of orthopedic trauma unit, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/1583
Record Dates: First submitted 2019-09-23; First posted 2019-09-27 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Proximal Humerus Fracture; 2 Part Fracture
Keywords: Proximal humerus fracture; Non-operative versus operative treatment; Conservative versus surgical treatment; Surgical versus non-surgical treatment
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 arms
Who Masked: Outcomes Assessor
Masking Description: The physiotherapists conducting outcomes at 6 months and 1 year do not know if patients are treated with surgery or not. Patients are instructed to wear t-shirt and not talk about treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical (No Intervention): No surgery
- Surgical (Active Comparator): Surgeons preference
  Interventions: Procedure: Open reduction internal stabilisation (ORIF)

INTERVENTIONS:
Procedure: Open reduction internal stabilisation (ORIF) — Treatment allocated to surgical or non-surgical group. Implant choice pragmatic, surgeons choice.
  Other Names: Surgery
  Arms: Surgical

SUMMARY:
The proximal humerus fracture (PHFs) is the third most common fracture type in the elderly, and represents 5% of the overall fractures. The incidence is increasing. The purpose of the project is to compare surgical and conservative management of two- part PHFs in light of radiological, economical and clinical outcome. Do the participants between 60 and 85 years of age with displaced two-part PHFs fare better or worse after surgery compared to non-operative treatment?

DETAILED DESCRIPTION:
The study-design is a single center single blinded randomized controlled trial (RCT) with 2 arms. Patients admitted to Akershus University Hospital (Ahus) with a displaced two-part proximal humeral fracture of OTA/ AO group 11A2 or 11A3 in need of surgical treatment will be randomly allocated to two groups; conservative/ non-operative treatment or open reduction and internal fixation (ORIF).

All following aims evaluated at controls at 6, 12, 26 and 52 weeks. The 6 months and 1 year controls will additionally be conducted by independent physiotherapists. The other controls are conducted by the treating surgeons. The physiotherapists will be blinded of chosen treatment, the patients wearing a t-shirt covering the shoulder at the consultations, hence single blinded RCT.

Primary aim: Functional outcome as evaluated by the Quick DASH (Disability of the arm, shoulder and hand) score at controls.

Preoperative evaluation:

The project participants will supervise and evaluate the data. General history, including; mechanism of injury, occupation, pre-existing medical conditions and medication, smoking history, American Society of Anesthesiologists Classification (ASA classification), BMI, hand dominance. At inclusion, the patient will be asked to fill out quick-Dash, Visual Analog scale (VAS), EQ-5D to determine the baseline-characteristics.

Postoperative evaluation:

Evaluation of postoperative radiographs for reduction of fracture and possible errors of the operative technique by the project participants and a radiologist.

Secondary aims:

1. Initial radiographic examination with standardized radiograph projections; true anterio-posterior projection and scapula projection pre- and post-operative. Registration of radiological complications defined by a reduction of Head-Shaft-Angle (HSA) of ≥10⁰ in frontal plane, screw penetration/cut-out, screw failure or failure of the osteosynthesis on radiographs. Evaluation of fracture healing/ non-union.
2. Evaluation of postoperative reduction: Reduction of tubercles, rotation of caput, re-establishment of medial support, position of calcar screws and distance from screws to cartilage in x-rays. Computer-tomographic scans are standard pre-operative practice at our institution. The problem of intra- and inter-observer reproducibility is a well-known confounder of fracture classification in proximal humeral fractures and CT scans will help clarify classification (19, 20) and fracture configuration. CT scan postoperatively will be taken within few days after surgery (Only in Stratum 1).
3. Qualitative Computed Tomography (QCT) is an alternative method to measure Bone Marrow Density (BMD) using a Hydroxyapatite plate/ a phantom. This is a flat plate placed under the shoulder during ordinary CT scanning. Several studies have demonstrated an association between the QCT measurements and risk of fragility fractures, so BMD will be assessed.
4. Functional outcome of surgical treatment as evaluated by Constant score by independent physiotherapists during follow-up. Measurement of strength according to recommendations given by the European Society of Shoulder and Elbow Surgeons ESSSE (http://secec.org/).
5. Functional outcome evaluated by Oxford Shoulder score, which is a validated patient-reported outcome measure. A shoulder-specific instrument designed to assess the outcome of all shoulder surgeries.
6. EQ-5D, a generic measure of health status that provide a simple descriptive profile used in clinical evaluation of health care. EQ-5D is recommended for use in cost-effectiveness in Health and Medicine and by the Washington panel of Pharmacoeconomics and outcomes research (ISPOR) task.
7. Health economic registration; length of hospital-stay, sick leaves, use of physiotherapy, appointments at general practitioners, extra controls at in-patient orthopedic clinic, removal of plate or nail, extra surgeries.
8. Monitoring complications such as deep or superficial infection, reoperations, avascular necrosis, non-union, nerve or vessel-damage.

In the literature, the following risk factors for failure of the osteosynthesis, Avascular necrosis (AVN) or chance of poor functional outcome are outlined; the factors will be examined as subgroups to see whether they are representative also for our population:

* A non-adequately reduced fracture. Evaluated in postoperative radiographs. Malalignment?
* Not adequately positioning of implant
* Degree of medial comminution and medial hinge (the amount of metaphyseal bone attached to the anatomic head fragment at trauma.
* Is sufficient medial support achieved in our patients, and if not, does the construction fail?
* Varus subsidence, measured as reduced Head shaft angle (HSA) (>10 degrees) during follow up
* Fixation in varus, HSA <120 or HSA <110 .
* Enough contact between head and shaft for healing?
* Age: Increasing age predisposes osteosynthesis failure and reduced function, probably because of decreasing bone density in proximal humerus in older age. The examiners want to examine whether there is a cut-off in age, in example 60, 65, 75, 80 or 85 years of age.
* Valgus >45 or Varus <30, which fracture is the worst?

Patients allocated to the conservative group may be offered surgical treatment if the fracture changes/ dislocates, in example no contact between the fracture ends if the patients activities of daily living (ADL) is greatly affected or pain is disproportionately

ELIGIBILITY:
-The study-design is a single center single blinded randomized controlled trial (RCT) with 3 arms. Patients admitted to Akershus University Hospital with a displaced 2-part proximal humeral fracture of OTA/ AO group 11A2 or 11A3 in need of surgical treatment will be randomly allocated to two groups; conservative/ non-operative treatment or open reduction and internal fixation (ORIF). The patients allocated to ORIF will be randomly allocated to either the Philos plate (Synthes) or the Multiloc nail (Synthes).

Inclusion criteria

1. Patients > 60 years and <85 years
2. More than 50% displacement between head or shaft or 50⁰ angulation of the head against the shaft in Y-projection or more than 45 ˚ valgus or more than 30˚ varus of the Head Shaft Angle (HSA).
3. Patient with tuberculum majus or minor fractures which displaced <5mm can be included as long as points 1 and 2 above are fulfilled.

Exclusion Criteria:

* Refusal to participate in the study
* Fracture more than 3 weeks old
* No contact btw head and shaft
* Ipsilateral damage that will influence the recovery and scoring systems
* Incapability to protect osteosynthesis, i.e. use of crutches because of injury to lower extremity. This is up to the treating surgeon to decide
* Pathological fracture or previous fracture of the same proximal humerus
* Multitrauma or "multifractured patient"
* Neurovascular injury
* Open fracture
* Noncompliance, dementia and/ or institutionalized
* Congenital anomaly
* Ongoing infectious process around the incision site for osteosynthesis
* Systemic disease that may influence healing processes or scoring systems (in example Rheumatoid arthritis/Multiple sclerosis/ poorly controlled DM)
* Fracture dislocation
* Substance abuse
* Inability to read and understand Norwegian
* Patients not residing in our catchment area
* Patients with a diameter of the humerus to small for nailing, will be allocated to the Philos-group.
* Any medical condition that excludes surgical treatment, including patients with ASA 3 or 4 that are considered too ill to go through surgery.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2034-10-31 (Estimated)

PRIMARY OUTCOMES:
Quick Dash | 1 year
  Prom, The QuickDASH is scored in two components: the disability/symptom section (11 items, scored 1-5) and the optional high performance sport/music or work modules (four items, scored 1-5). This is a 100-points scale where 0 is perfect/ best and 100 is the worst possible outcome

SECONDARY OUTCOMES:
Constant-Murley score | 1 year
  A clinical method of functional assessment of the shoulder, a 100-points scale composed of a number of individual parameters.
  >30 Poor 21-30 Fair 11-20 Good <11Excellent. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.
EQ5D | 1 year
  EQ-5D is a standardized instrument for measuring generic health status. The descriptive system element of the EQ-5D questionnaire produces a 5-digit health state profile that represents the level of reported problems on each of the five dimensions in EQ5D. EQ-5D health states may subsequently be converted into a single summary number, which reflects how good or bad a health state is according to the preferences of the general population of a country/region. EQ-5D is designed for self-completion. Further info and List of available value sets for the EQ-5D-3L:
  https://euroqol.org/docs/EQ-5D-3L-User-Guide.pdf
Radiology | 1 year
  Radiographs and CT scan before and after surgery, Radiographs of opposite shoulder for comparison
Number of patients with complications such as infection, Avascular necrosis, failure of osteosynthesis, screw cut out, nerve damage, deep vein thrombosis, | 1 year
  All complications registered; Infection, Avascular necrosis (AVN), osteosynthesis failure, screw cutout, varus of caput humeri, deep vein thrombosis
Visual Analog scale (VAS score) | 1 year
  VAS score for pain, a score designed for self-completion. The pain VAS is a unidimensional measure of pain intensity. The pain VAS is a continuous scale comprised of a horizontal line, 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme. The pain VAS is a single-item scale. "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100)

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn Aarøen, Professor, Study Director — Akershus Universitetssykehus HF
Locations (1):
- Akershus University Hospital, Lørenskog, Oslo County, Norway

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196